CLINICAL TRIAL: NCT01336166
Title: The Long-term Immunogenicity of an Inactivated Split-virion 2009 Pandemic Influenza A H1N1 Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SIBP-2009
Record Dates: First submitted 2011-04-07; First posted 2011-04-15 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2015-10

CONDITIONS: Influenza
Keywords: H1N1; Vaccine; Immunogenicity; Safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- split-virion, non-adjuvanted vaccine of 15 μg (Experimental): split-virion, non-adjuvanted H1N1 vaccine of 15 μg.
  Interventions: Biological: split-virion, non-adjuvanted H1N1 vaccine of 15 μg
- split-virion, non-adjuvanted vaccine of 30 μg (Experimental): split-virion, non-adjuvanted H1N1 vaccine of 30 μg.
  Interventions: Biological: split-virion, non-adjuvanted H1N1 vaccine of 30 μg
- split-virion, non-adjuvanted vaccine of 45 μg (Experimental): split-virion, non-adjuvanted H1N1 vaccine of 45 μg.
  Interventions: Biological: split-virion, non-adjuvanted H1N1 vaccine of 45 μg
- Placebo control (Placebo Comparator): Placebo control
  Interventions: Biological: Placebo control

INTERVENTIONS:
Biological: split-virion, non-adjuvanted H1N1 vaccine of 15 μg — 120 adults were assigned to receive 1 dose of 15μg split-virion, non-adjuvanted H1N1 vaccine.
  Arms: split-virion, non-adjuvanted vaccine of 15 μg
Biological: split-virion, non-adjuvanted H1N1 vaccine of 30 μg — 120 adults were assigned to receive 1 dose of 30μg split-virion, non-adjuvanted H1N1 vaccine.
  Arms: split-virion, non-adjuvanted vaccine of 30 μg
Biological: split-virion, non-adjuvanted H1N1 vaccine of 45 μg — 120 adults were assigned to receive 1 dose of 45μg split-virion, non-adjuvanted H1N1 vaccine.
  Arms: split-virion, non-adjuvanted vaccine of 45 μg
Biological: Placebo control — 120 adults were assigned to receive 1 dose of placebo.
  Arms: Placebo control

SUMMARY:
The aim of this study is to investigate the long-term immunogenicity and safety of the inactivated split-virion vaccine after one immunization.

ELIGIBILITY:
Inclusion Criteria:

1. Different age groups from 18 to 60 years, with normal intelligence and health. Volunteers (or their guardians) are well informed of the situation and sign the consent
2. Vaccination recipients qualified for this product have been inquired about medical history and clinically proven to be healthy
3. Requests of clinical research program can be obeyed
4. No other protective product is inoculated in last week
5. Axillary temperature below 37 degrees Celsius

Exclusion Criteria:

1. Volunteers in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination
2. Volunteers allergic to ingredient of vaccine composition (can be checked from vaccination history), especially to egg
3. History of progressive or severe neurologic disorder
4. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
5. Known or suspected impairment/alteration of immune function, for example receiving immunosuppressive therapy or receiving blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation
6. Asthma that is unstable or required emergent care, hospitalization or intubation during the past two years or that required the use of oral or intravenous corticosteroids
7. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
8. History of thyroidectomy or thyroid disease that required medication within the past 12 months
9. Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years
10. Guillain-Barre Syndrome
11. Self-reported seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C
12. Any other vaccines or immunoglobulin preparation within 1 weeks prior to enrollment
13. Axillary temperature ≥ 38.0 degrees Celsius within 3 days of intended study vaccination
14. Any conditions may influence the evaluation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Hemagglutination inhibition antibody titer | Day 180

SECONDARY OUTCOMES:
occurrence of solicited local and systemic adverse events after vaccination | Days 0-42

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial Center of Disease Prevention and Control, Changsha, Hunan, China